CLINICAL TRIAL: NCT00492154
Title: Fracture of Distal Radius and Ulna Healed With Shortening of One Bone. Clinical Significance at Skeletal Maturity
Status: Terminated | Type: Observational
Why Stopped: the study stopped because we could not recruit enough patients.
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Naum Simanovski, Hadassah Medical Organization
Other Study IDs: SIM04-HMO-CTILL
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-06

CONDITIONS: Forearm Injuries
Keywords: FRACTURE OF DISTAL RADIUS
MeSH Terms: conditions — Forearm Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The fractures of distal forearm are the most common trauma in children. Sometimes one of the bones becomes shortened as a result of fracture fragments overlap. When some amount of shortening exists, concern regarding relationship of distal radio-ulnar joint (DRUJ) arises. The common opinion is expressed in one of the textbooks and is represented by one sentence, which usually one bone shortening is well tolerated, probably does not cause a problem, and does not have clinical significance. However, pathology of ulna plus or minus variants is well described and may cause ulno-carpal abutting syndrome or radiocarpal pain. This concern may lead to more aggressive approach in treatment of a fracture, with attempts to make an equal bone length. We did not find in the literature study that investigates this problem. We postulate that obvious shortening of one bone may cause an inequality of DRUJ and can be clinically significant.

DETAILED DESCRIPTION:
We will evaluate the x-ray films of children that at the time of the injury were between the ages 1 day and 12 years. The selection of the x-ray films will be done based on the specific codes of the wrist x-rays (Ulna or Radius).

The evaluation will be merely to children that were treated in our hospital from 1996 to 2000.We are aiming to find cases when the fractures were healed with 1cm or more of shortening of one of the forearm's bones (Radius or Ulna).

We are going to compare these cases with another 20 patients with the same characteristics as the latter groups on the exception that their fractures were healed without shortening. The two groups will be matched by age, gender and the same diagnosis.

These patients will be summoned to the clinic when they are adult in respect to the skeletal maturity. The patients will be evaluated, including clinical examination of the hand wrists (left and right), motion rang, motor muscle function, description of abnormalities if there are and x-ray of both wrists.

ELIGIBILITY:
Inclusion Criteria:

* Children that had had Ulna or Radius X-rays
* Signing Informed consent.

Exclusion Criteria:

- Unwillingness to sign informed consent.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Boys and girls that are at lest 12 years old at the time of the wrist fracture.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-09

CONTACTS AND LOCATIONS:
Overall Officials: Naum Simanovski, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel